CLINICAL TRIAL: NCT05231070
Title: The Effect of Specialized Palliative Telemedicine for Patients with Advanced Cancer At Home
Brief Title: Specialized Palliative Telemedicine for Patients with Advanced Cancer
Acronym: TeleSPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Geana P Kurita, Senior Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R315A18018
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Cancer
Keywords: Cancer, telemedicine, dyadic coping, palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, in which patients will be randomly assigned either to one of the two arms (1:1): intervention (TeleSPC) or control group (standard care). Assessment will occur at inclusion (baseline) and after 2 weeks, 4 weeks, 8 weeks, and 6 months. sample will be composed by 87 patients in each group and their informal caregiver (1 informal caregiver per patient) .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TeleSPC (Experimental): Patients will be offered regular multidisciplinary video consultations with the SPC team and these patients and their informal caregiver will also be offered a dyadic psychological intervention.
  Regular multidisciplinary video consultations with multidisciplinary team, involvering cooperation between the section og Palliative medicine and the Department of Oncology, District nurse and the general practitioner.
  Operationel definition of informal caregiver: Patients will designated the closest person involved in their care (e.g., spouse, son/daughter, other relatives, and friends).
  Interventions: Other: TeleSPC
- Control (No Intervention): Patients will follow the current practice in the healthcare system (standard care). Control patients will be offered information to clarify the options available in case of unmet palliative needs. Patients' informal caregiver will be invited to participate in the study, but no intervention will be offered.

INTERVENTIONS:
Other: TeleSPC — Multidisciplinary video consultations with the SPC team. The team is multiprofessional and composed by physician, nurse, psychologist, social worker, physiotherapist and a chaplain, which is in line with the staffing of most SPC teams in Denmark and abroad. Video consultations will follow the same approach already used in physical consultations at the Section of Palliative Medicine, considering patients' changing needs and providing differentiated treatment and support, with the addition of a psychological intervention for dyadic coping between patient and closest informal caregiver
  Arms: TeleSPC

SUMMARY:
Specialized palliative care (SPC) plays an important role in providing patient-centered care and support to informal caregiver, besides establishing/intensifying/coordinating collaboration with primary and secondary health care sectors (hospital nurse/district nurse and general practitioner/oncologist) to improve care and support for patients and burdened informal caregiver. This study proposes to develop a SPC intervention enriched with a dyadic psychological intervention for patients with advanced cancer and their informal caregiver delivered by telemedicine at home (TeleSPC). It is our hypothesis that the intervention can enhance patient-centered care at home, support their informal caregiver, and improve relations/integration between the SPC teams, oncologic teams, the general practitioners and district nurses.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial in an open-label fashion, which proposes to develop a SPC intervention enriched with a dyadic psychological intervention (needs-based therapeutic framework based on existential-phenomenological therapy) for patients with advanced cancer and their informal caregiver delivered by telemedicine (video consultation) at home. The primary aim is to investigate the intervention effects on the patients' health-related quality of life (HRQoL). The secondary aims will be to analyze the intervention effects on number of hospitalizations, days spent at home, hospital admissions, survival, dyadic coping between patients and informal caregiver, staff satisfaction with the intervention and caregiver burden in patients' informal caregiver.

ELIGIBILITY:
Patient inclusion criteria:

* adults (at least 18 years old)
* solid organ cancer
* no longer receives curativ treatment
* provide written informed consent
* are able to speak and understand Danish Language
* are cognitively able to participate in the study
* have at least one symptom or problem with score ≥ 3 at the EORTC QLQ-C30

Patient exclusion criteria:

* primary brain cancer or central nervous system metastases
* a prognosis of less than six months
* incapable of cooperating in the trial
* already receive SPC

Informal caregiver inclusion criteria:

* adults (at least 18 years old)
* indicated by the patient as the closest informal caregiver
* able to speak and understand danish langues
* provide written informed consent

Informal caregiver exclusion criteria:

- refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline patient's health-related quality of life at 2 weeks, 4 weeks, 8 weeks, and 6 months | Baseline, 2 weeks, 4 weeks, 8 weeks, and 6 months
  The European Organisation for Research and Treatment of Cancer Quality of life Questionnaire - Core 30 (EORTC QLQ-C30) to assess several physical and psychosocial aspects of the patient's health-related quality of life. Scores range from 0 to 100; high values in the functioning and quality of life scales and low values in the symptoms scales indicate better outcomes.

SECONDARY OUTCOMES:
Change from baseline patients' use of health care system at 6 months | Baseline and 6 months
  Clinical information collected from patients' records regarding number of hospitalizations, days spent in hospital, and date of death
Change from baseline patients and informal caregiver dyadic coping at 4 weeks, 8 weeks, and 6 months | Baseline, 4 weeks, 8 weeks, and 6 months
  Dyadic Coping inventory to assess how patients and informal caregiver manage stress together concerning decision making and giving support to each other. Four subscales were selected to evaluate dyadic coping (dyad patient and relative/caregiver) regarding stress communicated by oneself (max. score 20), stress communication of the partner (max. score 20), common dyadic coping (max. score 25), and evaluation of dyadic coping (max score 10). Higher scores denote greater levels of the constructs measured by each subscale.
Change from baseline caregiver burden at 4 weeks, 8 weeks, and 6 months | Baseline, 4 weeks, 8 weeks, and 6 months
  Zarit Burden Interview to measure subjective burden among caregivers. Sum of scores ranges from 0 to 88. A score of 17 or more is considered high burden.
Change from baseline informal caregiver health related quality of life at 4 weeks, 8 weeks, and 6 months | Baseline, 4 weeks, 8 weeks, and 6 months
  RAND 36-Item Short Form Health Survey version 1.0. Scores range from 0 to 100; a higher score indicates a better result.
Healthcare professionals' satisfaction with intervention at 6 months | 6 months
  Interview with healthcare providers
Change from baseline patients' sleep at 2 weeks, 4 weeks, 8 weeks, and 6 months | Baseline, 2 weeks, 4 weeks, 8 weeks, and 6 months
  Pittsburg Sleep Quality Index to determining the quality and patterns of sleep. Global score ranges from 0 to 21; 0 indicates no difficult and 21 indicates severe difficlties in all areas.
Change from baseline patients' anxiety at 2 weeks, 4 weeks, 8 weeks, and 6 months | Baseline, 2 weeks, 4 weeks, 8 weeks, and 6 months
  Hospital anxiety and depression scale. Scores range from 0 to 21; 0-7 represent non-cases, 8-10 represent doubtful cases, and 11-21 represent definite cases.
Change from baseline patient's depression at 2 weeks, 4 weeks, 8 weeks, and 6 months | Baseline, 2 weeks, 4 weeks, 8 weeks, and 6 months
  Hospital anxiety and depression scale. Scores range from 0 to 21; 0-7 represent non-cases, 8-10 represent doubtful cases, and 11-21 represent definite cases.
Patients and informal caregivers' satisfaction with intervention at 6 months | 6 months
  Patients and informal caregivers will be requested to rate their satisfaction (scale 1-5), and will have the possibility to write any comment
Change from baseline informal caregivers' anxiety at 4 weeks, 8 weeks, and 6 months | Baseline, 4 weeks, 8 weeks, and 6 months
  Patient Health Questionnaires' scales (GAD-7). Seven items, each of which is scored 0 to 3, providing a 0 to 21 severity score.
Change from baseline informal caregivers' depression at 4 weeks, 8 weeks, and 6 months | Baseline, 4 weeks, 8 weeks, and 6 months
  Patient Health Questionnaires' scales (PHQ). Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Geana P Kurita, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, København Ø., Denmark

IPD SHARING:
Plan to Share IPD: No